CLINICAL TRIAL: NCT07075848
Title: Study of Outcomes of Delivery in Primgravida
Brief Title: Outcomes of Delivery in Primigravida
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salah Gobara, principal investigator, Assiut University
Other Study IDs: PGDA
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Vaginal Delivery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group
  Interventions: Procedure: vaginal delivery

INTERVENTIONS:
Procedure: vaginal delivery — follow up of progress of labour

SUMMARY:
Primigravida women are a high-priority population due to their increased risk of obstetric interventions and adverse outcomes compared to multiparous women. Research indicates that first-time mothers account for a disproportionate number of emergency cesarean sections and instrumental deliveries, often due to factors such as inadequate labor support or failure to progress

DETAILED DESCRIPTION:
The significance of auditing delivery care for primigravida women lies in their heightened vulnerability to complications such as prolonged labor, fetal distress, and higher rates of cesarean sections. Studies have shown that primigravida women often experience higher levels of fear and anxiety related to childbirth, which can influence their labor progression and overall birth experience. By systematically evaluating the care provided to this group, healthcare institutions can implement targeted interventions to enhance outcomes and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida women admitted for delivery at the hospital
* Singleton pregnancies.
* Gestational age ≥ 28 weeks (to exclude preterm deliveries before viability).
* Willingness to participate.

Exclusion Criteria:

* • Multiparous women.

  * Multiple pregnancies.
  * Women who decline to participate.
  * Deliveries occurring outside the specified study period.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primigravida come in labour
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
The rate of vaginal delivery in cases | 24 hours